CLINICAL TRIAL: NCT04160663
Title: Arterial Stiffness and Atrial Fibrillation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID and staffing issues study was terminated
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Hon-Chi Lee, M.D., Ph.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19-005443
Record Dates: First submitted 2019-10-31; First posted 2019-11-13 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Ultrasonography, Carotid Arteries

STUDY DESIGN:
Intervention Model Description: Carotid Ultrasound testing before and after a clinically scheduled cardioversion procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects with atrial fibrillation (Experimental): Subjects with atrial fibrillation that have been clinically scheduled for an electrical cardioversion procedure will have carotid ultrasound testing done before and after the procedure
  Interventions: Diagnostic Test: Carotid Ultrasound

INTERVENTIONS:
Diagnostic Test: Carotid Ultrasound — Uses sound waves to examine the blood flow through the carotid arteries and to determine the elastic properties or stiffness of the artery.

SUMMARY:
Researchers are trying to determine whether arterial stiffness detected by ultrasound can predict outcomes in the development and recurrence of atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* All patients with persistent AF, scheduled for electrical cardioversion

Exclusion Criteria:

* Unable to provide informed consent.
* Patients with intramural thrombus or other conditions that preclude the performance of electrical cardioversion.
* Patients with prior carotid stents.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-10-29 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-10-05 (Actual)

PRIMARY OUTCOMES:
Recurrence of Atrial Fibrillation following cardioversion | 6 months
  We will follow up by phone or look through medical records to record the number of subjects that have had a recurrence of Atrial Fibrillation. We are also looking if we can correlate the recurrence with arterial stiffness.

SECONDARY OUTCOMES:
Occurrence of heart failure | 6 months
  Number of subjects to have heart failure following cardioversion
Occurrence of stroke | 6 months
  Number of subjects to have a stroke following cardioversion
Occurrence of hospitalization | 6 months
  Number of subjects that have been hospitalized following cardioversion

CONTACTS AND LOCATIONS:
Overall Officials: Hon-Chi Lee, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials